CLINICAL TRIAL: NCT00936546
Title: A Protocol Based Treatment for Debilitating Fibrosing Skin Disorders With (Anti-CD 20), Rituximab, Evaluating Safety and Efficacy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/183
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Debilitating Fibrosing Skin Disorders (Localised Scleroderma, Eosinophilic Fasciitis)
MeSH Terms: conditions — Scleroderma, Localized; Eosinophilic Fasciitis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Mabthera, Rituximab 1000 mg I.V.

SUMMARY:
This study will evaluate the safety and efficacy of the combination of rituximab and methotrexate to treat disabling fibrosing skin disorders.Rituximab will be administered at baseline and month 6. The drug will be considered efficacious if the skin thickness diminishes substantially.

ELIGIBILITY:
Inclusion Criteria:

* (Fe) male >, = 18 years
* Fibrosing skin disorder, not fulfilling the ACR criteria for diffuse SSc
* Inadequate response to methotrexate (at least 12 weeks 10 mg/w, except if not tolerated or contra-indicated
* Debilitating disease defined by either one of the following:
* Restriction of mobility
* Disfiguration: eg: facial involvement
* Severe Internal Organ involvement
* Contraception for women with childbearing potential. Sexual abstinence is an alternative to contraception.

Exclusion Criteria:

* FVC<, = 50%
* LVEF<, = 40% of predicted value,
* DLCO<, = 40% of predicted value
* Exclusion criteria as specifically described in the protocol for anti-CD-20:
* Lack of peripheral venous access.
* Pregnancy or breast feeding.
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease).
* Evidence of significant uncontrolled concomitant disease such as, but not limited to, nervous system, renal, hepatic, endocrine or gastrointestinal disorders which, in the investigator's opinion, would preclude patient participation.
* Primary or secondary immunodeficiency (history of, or currently active), including known history of HIV infection.
* Known active infection of any kind (excluding fungal infections of mail beds), or any major episode of infection requiring hospitalization or treatment with i.v. anti-infectives within 4 weeks of baseline or completion of oral anti-infectives within 2 weeks prior to baseline.
* History of deep space/tissue infection (e.g. fasciitis, abscess, osteomyelitis) within 52 weeks prior to baseline.
* History of serious recurrent or chronic infection (for screening for a chest infection a chest radiograph will be performed at screening if not performed within 12 weeks prior to screening).
* History of cancer, including solid tumors, hematologic malignancies and carcinoma in situ (except basal cell and squamous cell carcinoma of the skin that have been excised and cured).
* History of a severe allergic or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of rituximab or to murine proteins.
* Concurrent treatment with any biologic agent or DMARD other than MTX. Treatment must be discontinued 14 days prior to baseline , except for the following: azathioprine for ≥ 28 days; leflunomide for ≥ 8 weeks (or ≥ 14 days after 11 days of standard cholestyramine or activated charcoal washout); infliximab ≥ 8 weeks; adalimumab ≥ weeks.
* Previous treatment with > 1 biological agent.
* Treatment with any investigational agent within 28 days of baseline or 5 half-lives of the investigational drug (which ever is the longer).
* Receipt of any vaccine within 28 days prior to baseline
* Intolerance or contraindications to i.v. glucocorticoids.
* Positive serum human chorionic gonadotropin (hCG) measured at screening or a positive pregnancy test prior to the first rituximab infusion.
* Positive tests for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C serology.
* Hemoglobin < 8.0 g/dL.
* Concentrations of serum IgG and/or IgM below 5.0 and 0.40 mg/mL, respectively.
* Absolute neutrophil count (ANC) < 1.5 X 10³/µL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-06; Primary Completion 2015-06-03 (Actual); Study Completion 2015-06-03 (Actual)

PRIMARY OUTCOMES:
Testing the safety of anti-CD-20 in a small cohort of patients with debilitating fibrosing skin disorders. | Safety will be evaluated at baseline, month 3, 6, 12, 15, 18, 24, 36, 48 and 60.

SECONDARY OUTCOMES:
Testing the efficacy of anti-CD-20 in a small cohort of patients with debilitating fibrosing skin disorders. | Efficacy will be evaluated at baseline, month 3, 6, 12, 15, 18, 24, 36, 48 and 60.

CONTACTS AND LOCATIONS:
Overall Officials: Filip De Keyser, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of the University Hospital Ghent — http://www.uzgent.be